CLINICAL TRIAL: NCT02627547
Title: Impact of Training Status of Endurance Athletes on Bioavailability of Flavanones
Brief Title: Impact of Training Status on Bioavailability of Flavanones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Senior Lecturer, University of Glasgow
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200120075
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Flavanones; Endurance-trained athletes; Biological availability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental tests (Experimental): 2 sets of experimental tests; once, during a period of normal training and repeated following one week of de-training
  Interventions: Behavioral: Normal training; Behavioral: De-training

INTERVENTIONS:
Behavioral: Normal training — 5-10 hours of endurance training each week
Behavioral: De-training — No training

SUMMARY:
Flavonoids are compounds that have been proven to have a beneficial effect on health, such as reducing the risk of developing cardiovascular disease and, in some cases, cancer. Citrus juices have a high flavonoid content. However, the absorption of flavonoids into the body is limited. This study will investigate whether being physically active improves the absorption of flavonoids.

Endurance trained athletes will be invited to participate. Following screening procedures (a. Health Screening Questionnaire; b. height and weight measurement for calculation of Body Mass Index; c. maximal oxygen consumption (VO2max) uptake test, eligible participants will undertake two experimental tests; one during a period of normal training, the other immediately following 1 week of detraining.

In the morning of the experimental trial participants will consume 500 mL of orange juice. Blood samples and urinary fractions will be collected prior (base line) to and for 24 hours after orange juice consumption. Participants will be asked to follow a special polyphenol-free diet and record weighed dietary intake for 2 days preceding each trial and during the day of the experimental trial.

The study aims to:

1. Determine the effects of training status of endurance athletes on bioavailability of flavanones in endurance trained individuals
2. Determine whether changes in bioavailability of flavanones are related to changes in biomarkers of inflammation, oxidative stress, plasma lipids and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* trained regularly for at least 4 years and typically perform at least 5 hours of endurance training per week (distance runners, triathletes, cyclists)
* healthy
* normotensive
* non-smokers
* not taking any drug therapies
* VO2 max >50 ml/kg body mass

Exclusion Criteria:

* history of gastrointestinal disease
* vegetarian
* unstable food habits
* VO2 max < 50 ml/kg body mass

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
• Plasma pharmacokinetics of naringenin, hesperetin, eriodictyol, isorhamnetin and phenolic acid metabolites | 24 hours
  Change in plasma concentrations collected at base line (0 hours) and 0.5,1, 2, 3,4,5,6,7,8, and 24 hours after ingestion of orange juice
• Urinary excretion of naringenin, hesperetin, eriodictyol, isorhamnetin and phenolic acid metabolites | 24 hours
  Change in concentrations in urinary fraction collected at base line (0 hours) and after ingestion of orange juice (0-5, 5-8, 8-10, 10-24 hours)

SECONDARY OUTCOMES:
Maximal Oxygen Consumption | 30 minutes
  Maximal Oxygen Consumption (ml/kg/min) measured in trained state by Douglas bag method
Body weight | 7 days
  Difference in body weight in kilograms between trained and detrained states measured by TANITA scales (TBF-300, Cranlea, UK)
Body fatness | 7 days
  Difference in percentage of body fat between trained and detrained states measured by bioelectrical impedance method (TBF-300, TANITA, Cranlea, UK)
Dietary Intake | 7 days
  Difference in energy/macronutrient intake between trained and detrained states measured from 7 day weighted food records

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Malkova, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow School of Medicine, Glasgow, United Kingdom

REFERENCES:
- [Derived] Pereira-Caro G, Clifford MN, Polyviou T, Ludwig IA, Alfheeaid H, Moreno-Rojas JM, Garcia AL, Malkova D, Crozier A. Plasma pharmacokinetics of (poly)phenol metabolites and catabolites after ingestion of orange juice by endurance trained men. Free Radic Biol Med. 2020 Nov 20;160:784-795. doi: 10.1016/j.freeradbiomed.2020.09.007. Epub 2020 Sep 11. PMID 32927016
- [Derived] Pereira-Caro G, Polyviou T, Ludwig IA, Nastase AM, Moreno-Rojas JM, Garcia AL, Malkova D, Crozier A. Bioavailability of orange juice (poly)phenols: the impact of short-term cessation of training by male endurance athletes. Am J Clin Nutr. 2017 Sep;106(3):791-800. doi: 10.3945/ajcn.116.149898. Epub 2017 Jul 26. PMID 28747329